CLINICAL TRIAL: NCT05195320
Title: Reinventing Yourself With Multiple Sclerosis (MS): An Intervention Aimed at Improving Self-Efficacy, Coping, Psychological Well-being, and Quality of Life in MS
Brief Title: Reinventing Yourself With Multiple Sclerosis (MS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: Craig Hospital (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-1164-21
Record Dates: First submitted 2021-11-15; First posted 2022-01-18 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A sample of 48 participants randomly assigned to either the intervention or control group (Intervention, N=24 and Controls, N=24) over four cohorts. Participants in each cohort will be randomized to either the intervention or control group with equal probability so that each group has 6 participants. That is, once 12 subjects have been recruited, they will form a cohort, be randomized into one of the two groups, and begin the study intervention; this process will continue until 48 subjects have been recruited into four cohorts.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Staff administering assessments will be blinded to group assignment (Intervention or control). Participants and group facilitators will be carefully instructed not to reveal group assignment to assessment administrators. Following each assessment, the blinded data collector will note whether unblinding occurred; this information will be entered into the study's web database. As an additional protection, blinded data collectors will have restricted access to the study database as some of the information that is collected would reveal group assignment (e.g., attendance of group members at sessions); this information will be entered into the database by unblinded staff. To track potential unblinding, blinded data collectors will respond to a two-item assessment of unblinding following each outcome assessment administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intervention (Experimental): Participants will attend six weekly two-hour facilitator-led sessions that include didactic presentations of eight core skills and related experiential exercises with extensive group discussion. These skills are presented in sequence over the course of the intervention so that participants can gain mastery of introductory concepts before undertaking those that are both more difficult and complex. The culmination of developing these skills and participation in a peer group will assist individuals in increasing self-efficacy and overall QOL, well-being and participation. Participants will complete follow-up assessment at 18- and 30-weeks post-intervention.
  Interventions: Behavioral: Reinvention with MS
- Placebo (Placebo Comparator): Participants will receive no intervention throughout the course of the study; however, the participants will be tested at 18- and 30-weeks participation in the study.
  Interventions: Behavioral: Reinvention with MS

INTERVENTIONS:
Behavioral: Reinvention with MS — A manualized group therapy to build self-efficacy among people living with multiple sclerosis.

SUMMARY:
Given the knowledge that detriments in QOL, well-being, and participation are common in MS and attributable in a large part to individual, person-specific factors (e.g., self-efficacy), efforts to develop interventions aimed at addressing these factors is well needed and likely to have a significant impact. The proposed investigation will consist of two phases involving participant recruitment and data collection. Phase 1 will consist of a focus group aimed at identifying the unique needs of individuals with MS, and findings will be used to adapt the Reinventing Yourself after Spinal Cord Injury (SCI) intervention to Reinventing Yourself with MS. Phase 2 will consist of a randomized controlled trial (RCT) in which the feasibility and efficacy of the intervention in a new population can be examined.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the leading cause of disability among middle-aged adults with recent estimates of nearly 1 million adults living with MS in the United States. Multiple sclerosis affects women anywhere from two to three times as often as men, with an age of diagnosis ranging from 20 to 50 years of age and a mean age of onset of 33 years of age. A host of physical, cognitive, and behavioral changes are common following the onset of this most common non-traumatic neurological disorder of middle adulthood, which greatly impacts quality of life (QOL), well-being, and everyday functioning and participation. Moreover, given that individuals are typically diagnosed with MS in the prime of their lives many are making important life decisions regarding work, family, etc. that are often hindered by their diagnosis. In fact, it has been found that men and women with MS aged 25-44, an age at which important early life decisions are often made, experienced more depression than their age-matched, healthy counterparts. Again, the course of the disease is variable and unpredictable with no known cure, which can lead to great uncertainty and difficulty in adjusting to a chronic and often, debilitating disease.

The overarching aim of the proposed investigation is to adapt the Reinventing Yourself intervention for use with MS and examine the feasibility and efficacy in increasing MS-specific and general self-efficacy and resilience, enhancing psychological well-being, fostering new ways of perceiving and managing one's illness in more proactive and positive ways, and improving participation in the community. To achieve this, the investigation has the following specific aims:

Specific Aim 1: Conduct a focus group with individuals with MS to identify unique needs of individuals with MS with regard to MS symptoms, barriers to well-being, QOL, and participation, and the role that person-specific factors (e.g., self-efficacy, resilience) and other psychological and social factors have contributed to success (or failure) in managing one's illness and living well.

Specific Aim 2: With the knowledge gained from Aim 1, modify the Reinventing Yourself intervention with the specific needs of MS, while maintaining the integrity and common principles of the Reinventing Yourself intervention.

Specific Aim 3: Conduct a RCT among individuals with MS to determine the feasibility and efficacy of the Reinventing Yourself with MS intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* 18 years of age or older
* English-speaking
* Able to provide informed consent
* Access to the internet (if needed should the groups have to be conducted online due to pandemic circumstances that may limit to in-person meetings).

Exclusion Criteria:

* History of any other neurological illness (e.g. traumatic brain injury, epilepsy, dementia)
* Cognitive impairment that would affect my ability to fully participate in the group
* (For in-person group): Live beyond a reasonable commuting distance (50+ miles)
* Any other medical or psychological condition that, in the judgement of the investigators, prevents successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Self-Efficacy Scale | Through study completion, an average of 6 months
  This scale measures self-efficacy related to the experience of MS symptoms and sequelae. Scores range from 14-84. Higher scores indicate greater self-efficacy.
General Self-Efficacy Scale | Through study completion, an average of 6 months
  This scale measures one's general ability to control their behaviors and execute goals. Scores range from 10-44. Higher scores indicate greater self-efficacy

SECONDARY OUTCOMES:
Health Status Questionnaire | Through study completion, an average of 6 months
  The Health Status Questionnaire consists for 8 scales: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Scores for each scale range from 0-100. Higher scores indicate less disability.
Satisfaction with Life Scale | Through study completion, an average of 6 months
  This scale measures global assessment of one's life on a scale of 5-35. Higher scores indicate greater satisfaction.
Ryff Psychological Well-being Scales | Through study completion, an average of 6 months
  This is a global assessment of quality of life. Scores range from 14-84. Higher scores indicate greater well-being.
Participation Assessment with Recombined Tools-Objective (PART-O) | Through study completion, an average of 6 months
  PART-O measures three domains of participation: Productivity; Social Relations; and Out and About. The short form consists of 17 items. Items are scored on a scale from 0 to 5, with higher scores indicating greater participation
Chicago Multiscale Depression Inventory | Through study completion, an average of 6 months
  This scale measures emotional distress among people with non-psychiatric medical illness across three scales: Mood, Evaluative, and Vegetative. 42 items are scored on a scale Higher scores indicate more negative affect.
State Trait Anxiety Scale | Through study completion, an average of 6 months
  This scale measures momentary (state anxiety) and general (trait anxiety). Scores range from 20-80. Higher scores indicate greater anxiety
Connor-Davidson Resilience Scale | Through study completion, an average of 6 months
  The Connor-Davidson Resilience scale (CD-RISC) measures stress-coping ability. The CD-RISC comprises of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience.
Benefit Finding in Multiple Sclerosis Scale | Through study completion, an average of 6 months
  This scale measures finding meaning and positive adjustment to MS. Scores range from 43-139. Higher scores indicate greater benefit finding.
Cope Inventory | Through study completion, an average of 6 months
  This instrument evaluates coping strategies. 28 items, scored from one ("I haven't been doing this at all") to four ("I've been doing this a lot"), exploring 14 strategies: active coping, planning, use of instrumental support, positive reframing, acceptance, use of emotional support, denial, venting, self-blame, humor, religion, self-distraction, substance use and behavioral disengagement. Higher scores reflect a higher tendency to implement the corresponding coping strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No